CLINICAL TRIAL: NCT06829537
Title: Study of the Prevalence of Endogenous Hypercortisolism in Patients With Resistant Hypertension in the United States of America (MOMENTUM)
Brief Title: Study of the Prevalence of Endogenous Hypercortisolism in Patients With Resistant Hypertension (MOMENTUM)
Acronym: MOMENTUM
Status: Recruiting | Type: Observational
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: Study 311
Record Dates: First submitted 2025-01-30; First posted 2025-02-17 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Resistant Hypertension; Hypercortisolism
Keywords: Hypercortisolism; Resistant Hypertension
MeSH Terms: conditions — Cushing Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a non-interventional study to assess the prevalence of endogenous hypercortisolism (eHC) in patients with resistant hypertension (rHTN) and will enroll approximately 1000 patients at approximately 45 sites in the United States (US).

Each patient will have an initial visit for screening. After eligibility is confirmed, a limited exam will be performed and demographic and medical history will be collected. Non-fasting labs and a urine collection will also be done. A second visit will be a fasting blood draw at 8 AM after taking 1 mg of dexamethasone the night before at 11 PM. Cortisol level and study labs will also be collected.

After the lab results are obtained, a third visit will be scheduled only for patients with eHC and will include a non-fasting blood draw at 8 AM and scheduling of a non-contrast CT scan.

DETAILED DESCRIPTION:
This is a non-interventional study enrolling approximately 1000 patients at approximately 45 sites in the (US) and will assess the prevalence of eHC in patients with rHTN.

For the purpose of this study, eHC is defined by post-dexamethasone suppression test (DST) cortisol > 1.8 μg/dL with serum dexamethasone levels ≥ 140 μg/dL in a population meeting the inclusion and exclusion criteria for this study.

rHTN is defined by the American Heart Association as 1) systolic blood pressure (SBP) above target (≥ 130 mmHg for purposes of this study) despite concurrent use of 3 or more antihypertensive medications from different classes including a diuretic at their maximally tolerated doses or 2) at target or above target SBP requiring concurrent use of 4 or more antihypertensive medications from different classes.

Each patient will have an initial visit for screening. After written informed consent and eligibility is confirmed including a urine pregnancy test (if applicable), blood pressure, weight, height and waist circumference will be checked, and medical history will be obtained. Non-fasting labs such as plasma renin activity, aldosterone, N-terminal-pro brain natriuretic peptide, complete blood count, high sensitivity C-reactive protein, hemoglobin A1c, and comprehensive metabolic panel will be collected. A urine test will also be performed for albumin to creatinine ratio.

A second visit will be at 8 AM (± 1 hour) the morning after taking 1 mg of dexamethasone at 11 PM the night before. The blood draw must be in the fasted state and will include cortisol level, lipid panel, adrenocorticotropic hormone (ACTH), and fasting glucose. Dexamethasone level will be checked automatically for any cortisol >1.8 μg/dL (eHC).

After the DST results are obtained, a third visit will be scheduled only for patients with eHC and will include a non-fasting 8 AM blood draw for ACTH and cortisol and scheduling of a non- contrast adrenal CT scan.

ELIGIBILITY:
Inclusion Criteria:

* Each patient must meet all of the following criteria to be enrolled in the study:
* Signed and dated Institutional Review Board (IRB)-approved informed consent form (ICF) prior to any study-specific screening procedures.
* Male/female patients must be 18 years or older at the time of signing the informed consent.
* Meet either of the following criteria:
* Has rHTN, defined by the American Heart Association as BP above target (systolic ≥ 130 mmHg for purposes of this study) despite concurrent use of 3 or more antihypertensive medications from different classes at their maximally tolerated doses, and 1 of these agents is a diuretic.
* Or, has rHTN, defined by the American Heart Association as SBP at target or above target requiring concurrent use of 4 or more antihypertensive medications of different classes.

Exclusion Criteria:

* Patients who meet any of the following criteria will not be permitted entry to the study:
* White coat hypertension, ie, elevated BP in the office only, as determined by the Investigator.
* Non-adherence to BP medications, as determined by the Investigator.
* Systemic glucocorticoid medications exposure (excluding inhalers or topical) within 3 months of screening. For temporary exposures to oral glucocorticoids the Medical Monitor may be consulted to determine eligibility.
* Has an historical estimated glomerular filtration rate (eGFR) < 30.
* Has severe untreated sleep apnea as determined by the Investigator.
* Has excessive alcohol consumption (eg, > 14 units/week for male, > 7 units/week for female) as determined by the Investigator.
* Has severe acute psychiatric, medical, or surgical illness, as determined by the Investigator.
* Is a woman who is pregnant or lactating. For women of childbearing potential, a urine pregnancy test must be negative before doing the DST. A woman of childbearing potential includes women < 50 years old, women whose surgical sterilization was performed < 6 months ago, and women who have had a menstrual period in the last 12 months.
* Is a woman who is on oral contraceptive pills (OCPs). Women on OCPs may be screened but must be willing and able to stop OCPs for at least 6 weeks prior to screening assessments. OCPs can be resumed immediately after the blood draw for the DST.
* Has history of congenital adrenal hyperplasia.
* Has had the diagnosis of Cushing syndrome and/or has used or plans to use any of the following treatments for Cushing syndrome:

  • Mifepristone, metyrapone, osilodrostat, ketoconazole, fluconazole, aminoglutethimide, etomidate, octreotide, lanreotide, pasireotide, longacting octreotide or pasireotide.
* Is unable to take dexamethasone due to a history of hypersensitivity or severe reaction to dexamethasone.
* Is a staff member working directly on the study or is a family member of someone working directly on the study, including any of the Sponsor's employees, the Investigator or the site staff.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Office-based care and university clinics in the United States.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-03-28 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
To assess the prevalence of endogenous hypercortisolism in a population with resistant hypertension. | From enrollment to the end of the study which is approximately 4 weeks.
  Prevalence of endogenous hypercortisolism in a population with resistant hypertension will be described as the percentage of patients with post-DST cortisol > 1.8 μg/dL with dexamethasone level ≥ 140 ng/dL among all patients enrolled.

SECONDARY OUTCOMES:
Assess clinical characteristics that increase the likelihood of a patient having endogenous hypercortisolism of those with and without abnormal adrenal imaging. | From enrollment to the end of the study which is approximately 4 weeks.
  - Clinical characteristics collected as medical history will be coded and presented by system organ class (SOC) and preferred term (PT).
Assess laboratory characteristics that increase the likelihood of a patient having endogenous hypercortisolism of those with and without abnormal adrenal imaging. | From enrollment to the end of the study which is approximately 4 weeks.
  Laboratory characteristics will be summarized using descriptive statistics (mean, standard deviation, minimum, maximum, and 95% CI for mean). All will be assessed to identify associations with endogenous hypercortisolism diagnosis.
Assess the likelihood of a patient having endogenous hypercortisolism of those with and without abnormal adrenal imaging. | From enrollment to the end of the study which is approximately 4 weeks.
  - In patients with endogenous hypercortisolism and resistant hypertension, the percentage of patients with and without abnormal adrenal imaging based on non-contrast CT scan.

CONTACTS AND LOCATIONS:
Locations (50):
- United States (50):
  - Site 378, Huntington Park, California
  - Site 406, La Jolla, California
  - Site 538, La Jolla, California
  - Site 041, Los Angeles, California
  - Site 535, Northridge, California
  - Site 379, Redondo Beach, California
  - Site 542, Santa Maria, California
  - Site 387, Tarzana, California
  - Site 375, Torrance, California
  - Site 533, Torrance, California
  - Site 553, Cooper City, Florida
  - Site 444, Edgewater, Florida
  - Site 528, Maitland, Florida
  - Site 554, Miami, Florida
  - Site 525, Miami, Florida
  - Site 527, Miami, Florida
  - Site 537, Port Charlotte, Florida
  - Site 009, Atlanta, Georgia
  - Site 552, Chicago, Illinois
  - Site 532, Winfield, Illinois
  - Site 046, Covington, Kentucky
  - Site 061, Metairie, Louisiana
  - Site 377, New Orleans, Louisiana
  - Site 410, Baltimore, Maryland
  - Site 394, Olney, Maryland
  - Site 440, Rockville, Maryland
  - Site 067, Boston, Massachusetts
  - Site 530, Troy, Michigan
  - Site 371, Las Vegas, Nevada
  - Site 541, Reno, Nevada
  - Site 070, Albany, New York
  - Site 524, New York, New York
  - Site 181, Chapel Hill, North Carolina
  - Site 536, Durham, North Carolina
  - Site 555, Greenville, North Carolina
  - Site 529, Mooresville, North Carolina
  - Site 540, Morrisville, North Carolina
  - Site 059, Wilmington, North Carolina
  - Site 436, Cincinnati, Ohio
  - Site 551, Cleveland, Ohio
  - Site 042, Cleveland, Ohio
  - Site 195, Columbus, Ohio
  - Site 168, Charleston, South Carolina
  - Site 534, Mt. Pleasant, South Carolina
  - Site 456, Austin, Texas
  - Site 370, Dallas, Texas
  - Site 526, Houston, Texas
  - Site 408, Lufkin, Texas
  - Site 369, San Antonio, Texas
  - Site 531, Weslaco, Texas

IPD SHARING:
Plan to Share IPD: Yes
Upon study completion, results will be presented at relevant scientific congresses and published in a peer-reviewed journal.